CLINICAL TRIAL: NCT03360461
Title: Intraoperative Imaging of Colon Cancer Using a Fluorescent Peptide (EMI-137) Against the c-Met Receptor
Brief Title: EMI-137 in Laparoscopic Colonic Resections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: Edinburgh Molecular Imaging Ltd (Unknown)
Responsible Party: Principal Investigator, David Jayne, Consultant Colorectal Surgeon, University of Leeds
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS16/87090
Record Dates: First submitted 2017-11-07; First posted 2017-12-04 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Colonic Cancer; Metastasis to Lymph Node
MeSH Terms: conditions — Colonic Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Intervention Model Description: Single-centre stage IIa developmental study, Open label, single arm, non-randomised feasibility study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EMI-137 (Experimental): Ten participants to receive the IMP - EMI-137 1 to 3 hours before laparoscopic colonic resection surgery. Dose range 0.02mg/kg to 0.13mg/kg will be administered.
  Interventions: Drug: EMI-137

INTERVENTIONS:
Drug: EMI-137 — EMI-137 - a fluorescent c-Met receptor targeted peptide

SUMMARY:
EMI-137 in laparoscopic colonic resections is a single-centre stage IIa developmental study.

Ten adult participants with a diagnosis of colon adenocarcinoma undergoing laparoscopic colonic will be recruited to the trial. Participants will receive a single intravenous dose of the IMP - EMI-137 1 to 3 hours before surgery. The ability of EMI-137 to produce visible intra-operative fluorescence of primary colon cancer and lymph node metastases will be explored and evaluated.

DETAILED DESCRIPTION:
EMI-137 in laparoscopic colonic resections is a single-centre stage IIa developmental study to explore and evaluate the ability of EMI-137 to produce visible intra-operative fluorescence of primary colon cancer and lymph node metastases.

The aim of this study is to investigate the ability of a fluorescent imaging agent - EMI-137 to produce visible fluorescence in colon cancer during laparoscopic surgery. EMI-137 consists of a cyanine dye coupled to a c-Met targeted peptide. It is supplied by Edinburgh Molecular Imaging Ltd. Colon cancer along with several other types of cancer over-express and/or show upregulation of the c-Met receptor. We anticipate, EMI-137 will accumulate in the tumour and any lymph nodes metastases when administered intravenously 1 to 3 hours before laparoscopic colonic resection surgery. The intravenous administration of EMI-137 may allow real-time intra-operative visualisation of colon cancer and any metastatic lymph nodes, aiding the safe and accurate resection of the tumour.

In total 10 patients will be recruited. Patients will have a diagnosis of primary colon adenocarcinoma, confirmed on biopsy or on radiological imaging, and will have been discussed at the colorectal cancer MDT meeting. Imaging will have been performed less than 8 weeks prior to surgery. Patients will be fit for surgical resection of the primary cancer. They may have suspected or confirmed distant metastatic disease. The planned procedure may be of palliative or curative intent. The anticipated recruitment period is six (6) months with one (1) month of trial follow-up.

Participants will receive written and verbal information, and allowed at least 24 hours to consider their participation in the trial. Participating patients will provide written, informed consent. Pre-operative patient demographics will be collected, including gender, age, BMI, baseline FBC, U&Es, LFTs and clotting profile, co-morbidities, ASA grade, and medication. All patients will undergo routine preoperative assessment, to include colonic imaging, and staging CT scan of chest, abdomen and pelvis. The planned procedure and radiological staging will be documented.

Patients will be administered an intravenous bolus of EMI-137 at a dose of between 0.02mg/kg to 0.13mg/kg EMI-137 2.5 hours (range 1 to 3 hours) prior to the surgical procedure start time (this refers to expected "knife to skin time"). The maximum dose will be 0.13mg/mg per patient for the total operative period. The time of administration will be recorded. Patients will be closely monitored for any adverse reactions to the medicinal product (as per schedule below).

The surgical procedure will be as per surgeon preference but must include laparoscopic surgery. The procedure must use a Near Infra-Red laparoscopic system such as the Karl Storz® endoscopic fluorescence imaging systems. It will be used to evaluate the colon cancer and regional lymph nodes under both white and red light. The presence of fluorescence within the primary cancer and any draining lymph nodes will be recorded relative to background fluorescence. The intensity of fluorescence will be recorded semi-quantitatively as: highly fluorescent, mildly fluorescent or isofluorescent to background. Mobilisation of structures to permit visualisation of the cancer and lymph nodes is permissible as long as the oncological principles of the operation are not compromised. Any fluorescent lymph nodes will be marked with a surgical clip (Ligaclip) to allow subsequent histopathological identification.

Postoperative care will be as routinely provided. Patients will be monitored for any adverse effects related to the medicinal product. Any adverse reactions as defined in the protocol below will be reported to the CI, clinical trial team, the industrial sponsor and where necessary, the appropriate regulatory bodies.

The histopathologists involved in the trial will examine the specimen using routine and trial specific histopathological techniques. The fluorescences obtained from the fresh frozen specimens will be appraised using the same semi-quantitative scale used intraoperatively; highly fluorescent, mildly fluorescent and isofluorescent. The tumour stage will be ascertained and compared against the pre-operative radiological stage. The degree of fluorescence obtained may also be compared against the level of c-Met expression and the morphological and functional characteristics of the tumour. Separate fresh tissue samples (unfixed cancer and normal mucosal tissue) will be taken, if accessible, and stored in a HTA-approved tissue bank.

Patients will be followed up as per routine practice. All patients will be reviewed in a colorectal clinic between 2 and 3 weeks following discharge, at which point their involvement in the study will cease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Patients with a diagnosis of colonic cancer (the disease can be of any radiological TMN stage and be located anywhere from the caecum up to but not including the rectosigmoid junction)
* Patients with or without distant visceral or lymphatic metastatic disease.
* Patients with synchronous colon cancers or polyps can participate.
* American Society of Anaesthesiologists (ASA) classification ≤3.
* Normal hepatic and renal function (eGFR ≥60 mls/min/1.73m2) and bilirubin within institutional limits and/or ALT ≤2.5x upper limit of institutional normal value) on serum laboratory blood tests performed ≤30 days prior to EMI-137 administration.
* Female participants who are surgically sterile (documented bilateral oophorectomy and/or hysterectomy), post-menopausal (cessation of menses for more than 1 year), or pre-menopausal with two negative urine pregnancy tests performed within 24 hours of administration of EMI-137 Injection.
* Pre-menopausal female participants of child-bearing potential who agree to employ two method of contraception (as defined in eligibility criteria of the protocol) during the study period and for 90 days after EMI-137 administration.
* Male participants with a non-pregnant female partner. Male participants with a pre-menopausal partner of child-bearing potential who agree to use two forms of contraception (as defined in section 8.2) during the study period and for at least 90 days after receiving EMI-137. (The only permissible exception would be if the participant had undergone documented bilateral orchidectomy or their female partner is post-menopausal (cessation menses >1 year) or has undergone documented bilateral oophorectomy and/or hysterectomy).

Exclusion Criteria:

* Patients who are participating in another intra-operative fluorescence study, or have participated in another fluorescence study within 3 months of the planned surgical procedure.
* Received an investigational medicinal product at any dose within 28 days of planned EMI-137 administration
* Patients with pre-existing inflammatory bowel disease.
* Patients who have undergone neoadjuvant chemotherapy to treat the colon cancer.
* Patients with impaired renal function (eGFR <60 mls/min/1.73m2).
* Patients with impaired liver function (Bilirubin above institutional limits and/or ALT >2.5x upper limit of normal).
* Pregnant and breastfeeding woman.
* Pre-menopausal woman planning to become pregnant within 90 days of receiving EMI-137; or pre-menopausal woman of child-bearing potential who refuse to use two forms of contraception for at least 90 days after receiving EMI-137.
* Male patients with a currently pregnant partner or male patients who are planning to conceive a pregnancy with a female partner within 90 days of receiving EMI-137; or male participants who refuse to use two forms of contraception as defined in section 8.2 for at least 90 days after receiving EMI-137 with their female partner of child-bearing potential.
* Poorly controlled or serious medical or psychiatric illness that, in the investigator's opinion, is likely to interfere with participation and/or compliance in this clinical trial.
* Previous adverse reaction to fluorescent agents.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-03-14 (Actual)

PRIMARY OUTCOMES:
To investigate the ability of EMI-137 to produce visible fluorescence in regional lymph nodes draining the colon cancer. | 6 months
  The ability of EMI-137 to detect colon cancer will be measured using the semi-quantitative descriptive terms of; highly fluorescent, mildly fluorescent and isofluorescent to background. The number of primary tumours highly or mildly fluorescent will be used to assess the success of EMI-137 as an imaging agent. The opinion of the senior operative surgeon performing the cases will also be taken in to consideration when appraising the efficacy of EMI-137.

SECONDARY OUTCOMES:
To investigate of the ability of EMI-137 to produce visible fluorescence in regional lymph nodes draining the colon cancer. | 6 months
  The ability of EMI-137 to detect metastatic lymph nodes will be measured using the semi-quantitative descriptive terms of; highly fluorescent, mildly fluorescent and isofluorescent to background. The number of lymph nodes deemed to be highly or mildly fluorescent intraoperatively will be used to measure the success of EMI-137 as an imaging agent. The opinion of the senior operative surgeon performing the cases will also be taken in to consideration when appraising the efficacy of EMI-137.
To investigate the concordance of visible fluorescence in colon cancer with histological stage and c-MET expression in resected specimens. | 6 months
  The resected specimen(s) will undergo thorough standard and trial-specific histopathological assessment. Cryosections will be taken from fresh frozen samples and analysed by fluorescent microscopy. The intraoperative fluorescence obtained will have been graded as either; highly fluorescent, mildly fluorescent or isofluorescent. The tumour stage will be ascertained and compared against the pre-operative radiological stage and the intraoperative fluorescence seen. High concordance will be a measure of success. The degree of fluorescence obtained may also be compared against the level of c-Met expression and the morphological and functional characteristics of the tumour. All comparisons will be made against the gold standard- standard histopathological assessment of the tumour, lymph nodes and the ascribed pathological stage of the tumour.
To investigate the concordance of visible fluorescence in cancer draining lymph nodes with histological evidence of metastasis. | 6 months
  The pre-operative predicted lymph node status will be compared against the pathological lymph node status and the intra-operative lymph node appearance with the administration of EMI-137. Step sectioning and cytokeratin staining of fluorescent nodes will be performed if metastatic disease is not identified during standard histopathological analysis. High concordance between the intraoperative appearance and the final TMN lymph node status will be used as a measure of success.
To explore the tumour (signal) to background (noise) florescence | 6 months
  The background (noise) appearance of nearby structures will be compared against the tumour and/lymph node (signal) in each case. High contrast between structures (high signal to noise ratio) will be used to measure the success of EMI-137 as an imaging agent. Factors likely to be negatively influencing the tumour to signal ratio will be evaluated and used to modify any further larger trials with EMI-137.
Investigation of the safety profile of EMI-137 | 7 months
  The number of adverse events (AE/AR/SAE/SUSAR) arising from the administration of EMI-137 or the related surgery will be measured and reported.
Exploration of systemic, operative, and patient factors, which adversely affect EMI-137 fluorescence detection of colon cancer. | 6 months
  Baseline demographic data will be analysed against the intraoperative and pathological results to determine any patient or surgical factors that negatively influence intra-operative visualisation with EMI-137. For example, Body Mass Index and tumour stage will be correlated to intraoperative results to determine possible adverse relationship.
Study of in vivo imaging compared against ex vivo fluorescent detection | 6 months
  8. Fluorescent microscopy of fresh frozen biopsies from the resected specimen will be analysed for fluorescence. This will be compared and contrasted against the intra-operative appearance of the tumour and draining lymph nodes with EMI-137. The results will compared against the gold standard - histopathological assessment of tumour characteristics and TMN (tumour, node and metastases) stage for concordance. High concordance will be used to measure the success of EMI-137 as an imaging agent.

CONTACTS AND LOCATIONS:
Locations (1):
- St James' University Hospital Trust, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Burggraaf J, Kamerling IM, Gordon PB, Schrier L, de Kam ML, Kales AJ, Bendiksen R, Indrevoll B, Bjerke RM, Moestue SA, Yazdanfar S, Langers AM, Swaerd-Nordmo M, Torheim G, Warren MV, Morreau H, Voorneveld PW, Buckle T, van Leeuwen FW, Odegardstuen LI, Dalsgaard GT, Healey A, Hardwick JC. Detection of colorectal polyps in humans using an intravenously administered fluorescent peptide targeted against c-Met. Nat Med. 2015 Aug;21(8):955-61. doi: 10.1038/nm.3641. Epub 2015 Jul 13. PMID 26168295